CLINICAL TRIAL: NCT03864146
Title: A Randomized Trial of Pioglitazone for the Treatment of Alcohol Use Disorder
Brief Title: Pioglitazone for the Treatment of Alcohol Use Disorder
Acronym: PAUSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NURA-015-18S; CX-001837-01 (Other Grant/Funding Number: Veterans Health CSR&D)
Record Dates: First submitted 2019-02-27; First posted 2019-03-06 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Alcohol dependence; Craving
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled parallel group study design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pioglitazone (Experimental): Pioglitazone titrated to 45mg by mouth each day
  Interventions: Behavioral: Brief Behavioral Compliance Enhancement Treatment
- Placebo (Placebo Comparator): placebo, identical 45mg pill
  Interventions: Behavioral: Brief Behavioral Compliance Enhancement Treatment

INTERVENTIONS:
Behavioral: Brief Behavioral Compliance Enhancement Treatment — This is a standardized 15-minute intervention that emphasizes medication adherence as a crucial element to change alcohol use behavior.
  Other Names: BBCET

SUMMARY:
Alcohol Use Disorder (AUD) is common among Veterans but medication treatment is used infrequently and the impact of these treatments are small to moderate at best. Pioglitazone, a medication FDA approved for diabetes, has been shown in pre-clinical studies to reduce alcohol. The proposed study will test the efficacy of pioglitazone to reduce alcohol use in a double-blind placebo controlled trial. Investigators plan to compare pioglitazone to placebo in 200 Veterans who have an AUD and who are currently drinking alcohol at two Veterans Affairs Health Care Centers. The primary hypothesis is that Veterans with an AUD who are currently drinking alcohol will have a greater reduction in alcohol use following treatment with pioglitazone compared to those treated with placebo.

DETAILED DESCRIPTION:
Background: Alcohol use disorder (AUD) and heavy drinking are common among Veterans with 42.2% of Veterans having a life-time history of AUD and 14.8% screening positive for past-year probable AUD. Although treatments for AUD have improved over the past several decades, more effective interventions are needed. Pioglitazone is an FDA approved medication used to treat diabetes. Pioglitazone is a PPAR agonist and has been reported to decrease voluntary alcohol consumption of a 10% alcohol solution in rats genetically selected for high alcohol consumption. In addition, when rats had to perform an operant task to receive alcohol, pioglitazone reduced alcohol self-administration but not saccharin intake. These data suggest that pioglitazone reduces the motivation to consume alcohol. No clinical studies of pioglitazone are available in patients with AUD only. This proposed research study is a double-blind controlled clinical trial of 200 Veterans with AUD randomized to either pioglitazone or placebo. The primary hypothesis is that Veterans with AUD who are currently drinking alcohol will have a greater reduction in heavy drinking days per week compared to those who receive placebo.

Methods: Male and Female Veterans who are above 18 years old, who are not seeking intensive outpatient alcohol treatment will be recruited from the Minneapolis and Long Beach VA Health Care Service's for the study. After screening visits and informed consent, participants who meet all inclusion and exclusion criteria and who sign the informed consent will be given a breathalyzer test and the following measures: The Structured Clinical Interview for DSM-5 (SCID), Obsessive Compulsive Drinking Scale (OCDS), Timeline Followback (TLFB), Beck Depression Inventory-2nd edition (BDI-II) and the PTSD Checklist (PCL-5). Participants will also provide a urine sample for a urine drug screen, Ethyl Glucuronide (EtG), and Ethyl Sulfate (EtS), and blood samples for ALT, AST and BNP (B-type natriuretic peptide). Women of childbearing potential will provide a urine sample for Beta-Human chorionic gonadotropin ( -HCG). Participants will then be randomized to receive either pioglitazone or placebo. The participants will be seen weekly for the first 4 weeks (visits 1,2,3,4- baseline or randomization visit will be visit 0) then every 2 weeks until the end of the study (week 6 or visit 5, week 8 or visit 6, week 10 or visit 7, week 12 or visit 8, and week 14 or visit 9) for a maximum of 12 visits (including the screening visit, baseline visit, and closeout visit). At week 16, there will be a termination or closeout visit after study medications have been tapered. During the first 2 weeks of the study, each subject will have their dose of pioglitazone (or placebo) increased to a dose of 45mg per day. In addition to the medication (pioglitazone or placebo all participants will receive Brief Behavioral Compliance Enhancement Treatment (BBCET) as their psychosocial treatment. This is a standardized 15-minute intervention that emphasizes medication adherence as a crucial element to change alcohol use behavior.

Alcohol use will be measured by the Timeline Follow-back method and biomarkers of alcohol use will also be measured to determine whether a reduction in alcohol correlates with reduced markers of alcohol use. In addition, the impact of pioglitazone on rumination and safety will be assessed with a variety of measures.

Relevance to Veterans Health: Veterans have high rates of AUD with significant impact on health, quality of life and mortality. In addition, the direct and indirect cost of AUD are high. Current medication treatment approaches are infrequently used and of only small to modest benefit. Pioglitazone has shown promise in several pre-clinical studies but no AUD clinically focused studies are available. If pioglitazone is found to be useful in reducing or eliminating alcohol use in Veterans it could be easily and rapidly repurposed to treat AUD, as it is already an FDA approved medication. Pioglitazone, given its unique mechanism of action, may offer an innovative approach to treating Veterans with AUD and thus help reduce the impact of this costly and difficult problem.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of at least moderate alcohol use disorder using the SCID
* A mean of six heavy drinking days per month for the 3-months prior to baseline.
* Drinking at least 14 drinks for men or 7 drinks for women, or more per week for the 4 weeks preceding the screening visit.
* Willingness to provide contact information to confirm study follow-up appointments
* Ability to perform informed consent
* Female subjects: a negative pregnancy test
* Serum ALT < 3 times reference range
* Stable psychiatric medication doses the month prior to baseline visit (antidepressant, antipsychotic, subjects may have changes in trazodone for sleep)

Exclusion Criteria:

* Current DSM-5 diagnosis of moderate to severe psychoactive substance use disorder (i.e. cocaine, opiates, methamphetamine) other than cannabis or nicotine
* Medical conditions contraindicating pioglitazone pharmacotherapy (e.g., congestive heart failure, clinically significant edema, clinically significant liver disease, hypoglycemia, diabetes, history of bladder cancer)
* Taking medications known to have significant drug interactions with the study medication (CYP2C8 inhibitors or inducers, antihyperglycemic medications)
* Cognitive or physical impairment that precludes study participation
* Currently and seriously suicidal (i.e., plan and intent)
* Currently being treated for AUD with a medication (naltrexone, naltrexone injectable, acamprosate, topiramate, disulfiram and gabapentin)
* Impending incarceration
* Pregnant or planning to become pregnant during the course of the trial or nursing for female patients
* Unwillingness to sign a written informed consent form
* Unwillingness to use a barrier method of birth control during the study for female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric W. Dieperink, MD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (2):
- United States (2):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant was randomized on July 26, 2019 and data were collected through March 29, 2024. Potential subjects were recruited from two VA medical centers (Long Beach and Minneapolis) and were recruited from outpatient mental health and medical clinics at each VA and through IRB approved advertisements. Also, a VA database was queried for all patients who scored greater than 3 on the AUDIT-C, recruitment letters were sent to a subset of these patients and recruited via this method.
Pre-assignment Details: Potential subjects who did not meet inclusion/exclusion criteria were not enrolled in the trial, this included 16 subjects who signed informed consent but did not meet criteria so a total of 185 subjects were randomized to drug
Period: Overall Study
Arm/Group | Pioglitazone | Placebo
Started | 93 | 92
Completed | 76 | 67
Not Completed | 17 | 25
Not completed — Lost to Follow-up | 14 | 23
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: Intent to treat analysis so all subjects were analyzed
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone | Placebo | Total
Number analyzed (Participants) | 93 | 92 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (14.1) | 51.5 (14.6) | 52.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 91 | 86 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 20 | 36
  White | 68 | 56 | 124
  More than one race | 1 | 6 | 7
  Unknown or Not Reported | 1 | 5 | 6
Baseline Characteristics [Count of Participants; unit: Participants] | 93 | 92 | 185

OUTCOME MEASURES:

1. Primary Outcome: Heavy Drinking Days Per Week Change
Description: The primary outcome is change in heavy drinking days per week as measured by the Timeline Follow-back. A heavy drinking day is defined as : >4 standard drinks in a day for men and >3 standard drinks in a day for women
Time Frame: Change between baseline and 14 weeks
Measure: Mean (95% Confidence Interval); unit: Mean heavy drinking days per week
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 93 | 92
Mean heavy drinking days per week | -1.76 [-2.37 to -1.14] | -2.3 [-2.94 to -1.66]

2. Secondary Outcome: Number of Subjects With no Heavy Drinking for the Last 8 Weeks of the Study
Description: The rate of no heavy drinking over the last 8 weeks of the study (weeks 6-14) is a responder analysis measure. This is the total count of participants of each group experiencing no heavy drinking days during weeks 7-14
Time Frame: heavy drinking between week 7 and 14
Population: The population of participants who were still in the study from weeks 7 through 14 were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 83 | 75
Participants | 51 | 49

3. Secondary Outcome: Number of Drinks Per Week
Description: Mean number of standard drinks per week as measured by the Timeline Follow-back
Time Frame: Change in mean drinks per week from baseline to week 14
Measure: Mean (95% Confidence Interval); unit: Change in mean drinks per week
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 93 | 92
Change in mean drinks per week | -20.15 [-27.3 to -13.0] | -21.20 [-28.6 to -13.8]

4. Secondary Outcome: Alcohol Craving
Description: Craving will be measured by the Obsessive Compulsive Drinking Scale (OCDS). Range is 0-56, greater scores indicates greater craving.
Time Frame: Change in mean obsessive compulsive drinking scale score from baseline to week 14
Measure: Mean (95% Confidence Interval); unit: Total OCDS score
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 93 | 92
Total OCDS score | -5.30 [-6.37 to -1.63] | -4.0 [-7.76 to -2.84]

5. Secondary Outcome: Ethyl Glucuronide (EtG) and Ethyl Sulfate (EtS) Positivity
Description: EtG and EtS are direct metabolites of alcohol and remains in urine for up to 5 days after cessation from alcohol and they are highly sensitive with good specificity for alcohol use. ETG and ETS results are dichotomous and scored as either positive or negative for alcohol.
Time Frame: Change between baseline and 14 weeks
Measure: Mean (95% Confidence Interval); unit: change in ETG/ETS positive tests
Arm/Group | Pioglitazone | Placebo
Number analyzed (Participants) | 93 | 92
change in ETG/ETS positive tests | 0.00 [-0.178 to 0.178] | -0.03 [-0.219 to 0.154]

ADVERSE EVENTS:
Time Frame: 14 weeks (baseline to week 14)
Description: Adverse events were gathered from a checklist developed for the study based on adverse events from pioglitazone package insert. Subjects may be affected by more than one adverse event.
Arm/Group | Pioglitazone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/92
Serious Adverse Events (participants affected / at risk) | 5/93 | 6/92
Other Adverse Events (participants affected / at risk) | 76/93 | 76/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=93) | Placebo (N=92)
Alcohol intoxication (Psychiatric disorders) | 3 (9) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
chest pain (Cardiac disorders) | 1 (1) | 0 (0)
gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pioglitazone (N=93) | Placebo (N=92)
Edema (Blood and lymphatic system disorders) | 24 (68) | 21 (48)
Weight gain (General disorders) | 29 (42) | 18 (34)
Cough (Respiratory, thoracic and mediastinal disorders) | 50 (114) | 36 (80)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 44 (96) | 39 (101)
Muscle pain (Musculoskeletal and connective tissue disorders) | 32 (80) | 32 (67)
Fatigue (General disorders) | 48 (100) | 46 (99)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 29 (48) | 19 (29)
Blurred vision (Eye disorders) | 29 (64) | 30 (53)
Nausea (Gastrointestinal disorders) | 7 (7) | 9 (9)
Headache (General disorders) | 7 (8) | 5 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT03864146/Prot_SAP_001.pdf
  • Informed Consent Form (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT03864146/ICF_000.pdf